CLINICAL TRIAL: NCT03072602
Title: A Study of Racial Differences in Natriuretic Peptides Response to Glucose Challenge
Brief Title: Racial Differences in the Natriuretic Peptide Response to Glucose Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pankaj Arora, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: X16081002
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy; Natriuretic Peptides; Metabolic Syndrome
Keywords: Racial differences
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Each participant will be enrolled into one of the two groups by race.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- African-American (Experimental): Healthy self-identified African-American participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB). On 4th day, participants will come to the clinic in fasting state and drink 75 gm of oral glucose solution, followed by blood collection every hour for 8 hours.
  Interventions: Dietary Supplement: Study diet; Other: Glucose Challenge
- White (Active Comparator): Healthy self-identified white participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB). On 4th day, participants will come to the clinic in fasting state and drink 75 gm of oral glucose solution, followed by blood collection every hour for 8 hours.
  Interventions: Dietary Supplement: Study diet; Other: Glucose Challenge

INTERVENTIONS:
Dietary Supplement: Study diet — Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB).
Other: Glucose Challenge — Participants will come in fasting state on the main study visit day and will be given 75 gm oral glucose solution to drink, followed by blood collection every hour for next 8 hours.

SUMMARY:
The purpose of the study is to discover any racial dissimilarity in the response of Natriuretic peptide (NP) system to acute metabolic influences such as a high carbohydrate challenge

DETAILED DESCRIPTION:
Previous studies have shown an association between reduced levels of circulating natriuretic peptides (NPs) and obesity in humans. This association is especially pronounced in those with metabolic syndrome traits and elevated plasma insulin. As previously conducted study has shown that an increase in NPs with weight loss in obese individuals is "primary" and not secondary to alteration in cardiac structure or function.

Previous experimental data suggests that Atrial NP (ANP) has a wide range of favorable metabolic effects including that activation of brown fat and improvement in skeletal muscle oxidative capacity and glucose utilization. New evidence suggests that ANP activation directly modulates insulin sensitivity and energy homeostasis, suggesting that ANP suppression could promote more obesity/insulin resistance. Moreover, ANP exerts potent lipolytic effects in vitro and in vivo. The previous study has shown that a high-carbohydrate challenge in healthy volunteers is associated with a reduction in N-terminal-proANP (NTproANP) but not N-terminal-proB-type NP (NTproBNP) levels. Nonetheless our outcomes were predominantly in Caucasians and warrants replication in other racial groups.

There is no data on the ANP response to high-carbohydrate challenge in African Americans, a racial group with disproportionately greater rates of obesity, insulin resistance, and diabetes as compared to Caucasians. So the investigators have proposed to conduct a pilot study in otherwise healthy, normotensive subjects to examine NP system, especially the effects on MRproANP in response of high-carbohydrate challenge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Blood pressure less than 140/90
* Estimated creatinine clearance >60cc/min
* Willingness to comply with the study diet

Exclusion Criteria:

* History of hypertension
* History of cardiovascular, renal, or liver disease
* Diabetes or use of glucose-lowering medications
* Use of vasoactive or diuretic medications
* Atrial fibrillation
* Anemia (Hematocrit < 41% in men and <35% in women
* Abnormal serum sodium or potassium
* Urine β-HCG consistent with pregnancy
* Abnormal liver function tests (>3x upper limit of normal)
* Women taking hormonal birth control
* Current smokers
* Regular users of non-steroid anti-inflammatory medications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Arora, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora P, Wu C, Hamid T, Arora G, Agha O, Allen K, Tainsh RET, Hu D, Ryan RA, Domian IJ, Buys ES, Bloch DB, Prabhu SD, Bloch KD, Newton-Cheh C, Wang TJ. Acute Metabolic Influences on the Natriuretic Peptide System in Humans. J Am Coll Cardiol. 2016 Feb 23;67(7):804-812. doi: 10.1016/j.jacc.2015.11.049. PMID 26892417
- [Background] Arora P, Reingold J, Baggish A, Guanaga DP, Wu C, Ghorbani A, Song Y, Chen-Tournaux A, Khan AM, Tainsh LT, Buys ES, Williams JS, Heublein DM, Burnett JC, Semigran MJ, Bloch KD, Scherrer-Crosbie M, Newton-Cheh C, Kaplan LM, Wang TJ. Weight loss, saline loading, and the natriuretic peptide system. J Am Heart Assoc. 2015 Jan 16;4(1):e001265. doi: 10.1161/JAHA.114.001265. PMID 25595796
- [Background] Wu C, Arora P, Agha O, Hurst LA, Allen K, Nathan DI, Hu D, Jiramongkolchai P, Smith JG, Melander O, Trenson S, Janssens SP, Domian I, Wang TJ, Bloch KD, Buys ES, Bloch DB, Newton-Cheh C. Novel MicroRNA Regulators of Atrial Natriuretic Peptide Production. Mol Cell Biol. 2016 Jun 29;36(14):1977-87. doi: 10.1128/MCB.01114-15. Print 2016 Jul 15. PMID 27185878
- [Result] Patel N, Russell GK, Musunuru K, Gutierrez OM, Halade G, Kain V, Lv W, Prabhu SD, Margulies KB, Cappola TP, Arora G, Wang TJ, Arora P. Race, Natriuretic Peptides, and High-Carbohydrate Challenge: A Clinical Trial. Circ Res. 2019 Nov 8;125(11):957-968. doi: 10.1161/CIRCRESAHA.119.315026. Epub 2019 Oct 6. PMID 31588864

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 81 participants agreed to participate in the study following the completion of the informed consent process and were assigned to each Arm/group. We had 7 study dropouts and 2 participants were not able to complete the protocol. A total of 72 participants completed the study.
Groups:
- African American: Healthy self-identified African American participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB). On the 4th day, participants will come to the clinic in a fasting state and drink 75 gm of oral glucose solution, followed by blood collection every hour for 8 hours.
  Study diet: Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB).
  Glucose Challenge: Participants will come in a fasting state on the main study visit day and will be given 75 gm oral glucose solution to drink, followed by blood collection every hour for the next 8 hours.
- White: Healthy self-identified White participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB). On the 4th day, participants will come to the clinic in a fasting state and drink 75 gm of oral glucose solution, followed by blood collection every hour for 8 hours.
  Study diet: Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB).
  Glucose Challenge: Participants will come in a fasting state on the main study visit day and will be given 75 gm oral glucose solution to drink, followed by blood collection every hour for the next 8 hours.
Period: Overall Study
Arm/Group | African American | White
Started (81 participants started the study; 39 Blacks and 42 Whites) | 39 | 42
Total Participant Screened for the Purpose of Eligibilty (94 participants were screened for eligibility) | 47 | 47
Ineligible Participants (13 determined ineligible by screening labs) | 8 | 5
Participant Received Standardized Meals (81 Participants received 3 days of standardized meals to control for salt intake) | 39 | 42
Study Dropouts (7 study dropouts) | 4 | 3
Participants Returned for Glucose Challenge Protocol (74 participants returned for the glucose challenge protocol) | 35 | 39
Unable to Complete the Protocol | 1 | 1
Completed (72 participants completed the study; 34 Blacks and 38 Whites) | 34 | 38
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African-American | White | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Customized [Median (Inter-Quartile Range); unit: years] | 27 [21 to 33] | 26 [22 to 30] | 27 [21 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 0 | 34
  White | 0 | 38 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [24 to 31] | 25 [22 to 27] | 26 [22 to 31]
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mmHg] | 115 [108 to 124] | 112 [105 to 118] | 114 [105 to 124]
Sodium [Median (Inter-Quartile Range); unit: mmol/L] | 139 [138 to 140] | 139 [137 to 140] | 139 [137 to 140]
Potassium [Median (Inter-Quartile Range); unit: mmol/L] | 4.0 [3.9 to 4.3] | 4.1 [3.9 to 4.3] | 4.1 [3.9 to 4.3]
Creatinine [Median (Inter-Quartile Range); unit: mmol/L] | 0.8 [0.8 to 1.0] | 0.8 [0.7 to 1.0] | 0.8 [0.7 to 1.0]
Percentage of Hematocrit [Median (Inter-Quartile Range); unit: %] | 40 [37 to 43] | 40 [39 to 43] | 40 [37 to 43]
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 93.7 (11.6) | 93.1 (5.8) | 93.4 (9.0)
Fasting Insulin [Mean (Standard Deviation); unit: mg/dL] | 14.3 (18.4) | 6.6 (3.6) | 10.2 (13.4)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: Ratio] — HOMA-IR is used to estimate insulin resistance. HOMA-IR = Fasting insulin levels in mU/l X Fasting glucose levels in mg/dl/405. The normal HOMA-IR value in healthy humans ranges from 0.5-1.4. The HOMA-IR value greater than 2.5 indicates significant insulin resistance. The HOMA-IR above 1.9 indicates early insulin resistance.
  Ratio | 3.6 (5.8) | 1.5 (0.9) | 2.5 (4.2)
Mid-regional pro-atrial natriuretic peptide (MRproANP) [Median (Inter-Quartile Range); unit: pmol/L] | 43 [33 to 55] | 52 [45 to 65] | 48 [33 to 65]
B-type natriuretic peptide (BNP) [Median (Inter-Quartile Range); unit: pg/mL] | 17 [13 to 23] | 22 [18 to 33] | 20 [13 to 33]
N-terminal pro-B-type natriuretic peptide (NTproBNP) [Median (Inter-Quartile Range); unit: pg/mL] | 14 [14 to 23] | 33 [18 to 53] | 24 [14 to 53]

OUTCOME MEASURES:

1. Primary Outcome: Plasma MRproANP
Description: Change in circulating MRproANP levels in response to glucose challenge in African-Americans (Linear mixed models using MRproANP as the dependent variable and time as the independent variable were used. Values are predicted log MRproANP with 95% CI)
Time Frame: From 1st hour to 10th hour on the main study visit day after consuming study meals for 3 days
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | African-American
Number analyzed (Participants) | 34
Percentage of change | 23 [19 to 27]

2. Secondary Outcome: The Difference in Circulating Plasma MRproANP
Description: Change in circulating MRproANP levels in response to glucose challenge between African-Americans and whites (Linear mixed models using MRproANP as the dependent variable and time as the independent variable were used. Values are predicted log MRproANP with 95% CI)
Time Frame: From 1st hour to 10th hour on the main study visit day after consuming study meals for 3 days
Measure: Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Whites: Healthy self-identified white participants will be enrolled and each will undergo a physical exam and screening tests to determine participants' eligibility. Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB). On 4th day, participants will come to the clinic in fasting state and drink 75 gm of oral glucose solution, followed by blood collection every hour for 8 hours.
  Study diet: Participants will consume the study diet for 3 days provided by the clinical research unit's metabolic kitchen (at UAB).
  Glucose Challenge: Participants will come in fasting state on the main study visit day and will be given 75 gm oral glucose solution to drink, followed by blood collection every hour for next 8 hours.
Arm/Group | African-American | Whites
Number analyzed (Participants) | 34 | 38
Percentage change | 23 [19 to 27] | 34 [31 to 38]

3. Secondary Outcome: Serum Insulin
Description: The difference in serum insulin levels at 1 hour in response to glucose challenge between African-Americans and whites
Time Frame: At 1 hour after glucose challenge
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | African-American | Whites
Number analyzed (Participants) | 34 | 38
µU/mL | 98.5 (10.1) | 69.7 (6.7)

4. Secondary Outcome: Serum Glucose
Description: The difference in serum glucose levels at 1 hour in response to glucose challenge between African-Americans and whites
Time Frame: At 1 hour after glucose challenge
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | African-American | Whites
Number analyzed (Participants) | 34 | 38
mg/dL | 129.9 (7.3) | 126.8 (6.2)

5. Secondary Outcome: Plasma NTproBNP
Description: Change in circulating NTproBNP levels in response to glucose challenge in African-Americans and Whites (Linear mixed models using MRproANP as the dependent variable and time as the independent variable were used. Values are predicted log NTproBNP with 95% CI)
Time Frame: From 1st hour to 10th hour on the main study visit day after consuming study meals for 3 days
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | African-American | Whites
Number analyzed (Participants) | 34 | 38
Percentage | -1 (0.2) | -3 (0.3)

6. Secondary Outcome: Change in Neprilysin (Membrane Metalloendopeptidase) mRNA Expression Levels Between African-Americans and Whites
Description: The relative circulating Neprilysin (Membrane Metalloendopeptidase) mRNA quantification (fold change) at baseline between African-Americans and Whites
Time Frame: At baseline
Measure: Mean (Standard Error); unit: fold change
Arm/Group | African American | White
Number analyzed (Participants) | 20 | 29
fold change | 3.4 (0.79) | 1.0 (0.15)

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | African American | White
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 0/34 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03072602/Prot_SAP_001.pdf
  • Informed Consent Form (2019-07-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03072602/ICF_000.pdf